CLINICAL TRIAL: NCT06292260
Title: Multi-functional Innovative Digital Toolkit for the Skin Diseases n LMICs and Beyond
Brief Title: Digital Toolkit for Skin Diseases in LMICs: Part 2
Acronym: MIND-the-SKIN2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Hope Commission International (Unknown); Institut Pasteur of Cote d'Ivoire (Other Government); Institut Raoul Follereau (Unknown); Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other); Tokyo Medical and Dental University (Other)
Responsible Party: Principal Investigator, Rie Yotsu, Associate Professor, Tulane University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-2054-2
Record Dates: First submitted 2024-02-23; First posted 2024-03-05 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Skin Diseases
Keywords: Skin Diseases; Neglected Diseases; Teledermatology; Telemedicine; Remote Consultation
MeSH Terms: conditions — Skin Diseases; Neglected Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- With mHealth app (Experimental): All healthcare providers will receive the mHealth app (eSkinHealth) to be used in their daily practices.
  Interventions: Device: mHealth app

INTERVENTIONS:
Device: mHealth app — The eSkinHealth app is a tablet application that can be used as a portable patient chart for dermatological conditions in areas with poor internet connectivity, and for teledermatology when in need.

SUMMARY:
Impact evaluation of eSkinHealth in improving case detection of skin NTDs and treatment outcomes in rural and urban settings

DETAILED DESCRIPTION:
A key component of integrated community-based surveillance using the digital health tool is to boost case detection for skin NTDs in the co-endemic target regions as well as to support follow-up management of those cases detected. The project uses the 'eSkinHealth' app which the investigators developed. The application offers a platform for facilitating field-based screening by community health workers (CHWs) and assisting primary healthcare workers (PHWs) (i.e., nurses in the case of Côte d'Ivoire) in remote diagnosis and case management through teledermatology involving specialized dermatologist. Upon consultation, identification and demographic data will be collected from an individual with suspected lesions and photos of skin lesions will be taken and uploaded in the patient files. These will then be cross-checked by remote dermatologists to confirm the clinical diagnosis and facilitate referral of identified cases to the health facility for early initiation of treatment. When patients are enrolled for treatment, regular remote dermatological consultations are expected to improve the follow-up and ensure better treatment outcomes.

For the evaluation of eSkinHealth app performance for this study, comparison will be made on the impact of having the app between rural and urban settings. This approach will allow the assessment whether the system is useful and expandable to a wider region of Côte d'Ivoire. The evaluation will be performed with focus on skin NTDs (such as Buruli ulcer, leprosy, mycetoma, lymphatic filariasis, scabies, and yaws) as the target diseases as these are chronic conditions with well-described disease course.

A total of 48 PHWs from two health districts of Abidjan will be selected. They will be compared against the 48 PHWs from Sinfra and Bouaflé health districts who had been a part of the previous study.

Trainings on eSkinHealth app, dermatological photography, and skin NTDs and basic dermatology will be provided to our participants. Patients with skin lesions will be asked to be part of the study and will be registered in the eSkinHealth app upon informed consent. Remote dermatologists will be recruited on a voluntary basis. Diagnosed cases will be managed and followed up as per national guidelines for each disease.

ELIGIBILITY:
1. Healthcare providers (i.e., doctors, nurses, or community health workers/volunteers)

   Inclusion Criteria:
   * 18 years or older
   * Working at primary health centers or clinics in Cote d'Ivoire
   * Able to read and speak fluent French
   * Willing to participate in the pilot study for the 12-month study duration
   * Willing to use a provided tablet with the eSkinHealth app if they were assigned to the intervention group
   * Able to consent for oneself

   Exclusion Criteria:
   * Planning to leave their job at the clinics within the study period
   * Difficulty operating mobile devices
2. Patients with skin diseases

Inclusion Criteria:

* Clinically suspected or diagnosed with skin NTDs (Buruli ulcer, leprosy, and yaws) or have other clinically diagnosed skin conditions
* Able to consent for oneself

Exclusion Criteria:

* Clinically diagnosed skin conditions outside of the target site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of cases of each skin NTD (neglected tropical disease) and other skin conditions as compared to the pre-intervention | 12 months
  Differences in case numbers diagnosed and followed up between the rural and urban areas. The case numbers will be retrieved from the eSkinHealth server registry which data will be exported to Excel for analysis.

SECONDARY OUTCOMES:
Case confirmation rate for each skin NTD (neglected tropical disease) and other skin conditions by dermatologists | 12 months
  Case confirmation data by dermatologists will be retrieved from the eSkinHealth server registry which data will be exported to Excel for analysis.
Number of days from registry to confirmatory diagnosis | 12 months
  Dates of registry and diagnosis will be retrieved from the eSkinHealth server registry which data will be exported to Excel for analysis.
Feasibility, usability, and effectiveness of the surveillance approach using eSkinHealth app | 12 months
  This will be evaluated using the System Usability Scale (SUS) tool and semi-structured in-depth interviews.
Capacity building and effectiveness of training | 12 months
  This will be evaluated using the pre- and post-test results and by diagnostic accuracy by primary health workers (PHWs) over time measured through the eSkinHealth server registry.

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Commission International, Abidjan, Côte d’Ivoire